CLINICAL TRIAL: NCT06180239
Title: Different Segmentectomy vs Lobectomy Comparison in NSCLC
Brief Title: Segmentectomy vs Lobectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Regina Elena Cancer Institute (Other); Istituto Europeo di Oncologia (Other); University of Pisa (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Principal Investigator, CHIAPPETTA MARCO, Dr, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6146
Record Dates: First submitted 2023-12-04; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer Stage I; Surgery
Keywords: segmentectomy; lobectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Single Segmentectomy group: patients underwent single segment resection,
- Lobectomy group: Patients underwent lobectomy
- Multiple segmentectomy group: patients underwent multiple segments resection,

SUMMARY:
Actual indications for stage Ia NSCLC patients suggest lobectomy and lymphadenectomy. On the other hand, recent studies reported non-inferiority of segmentectomy in case of nodule < 2cm or with ground glass appearance at computed tomography.

However, most of these studies did not report specifical analysis on kind of segmentectomy (single or multiple) and kind of lobectomy. Moreover, a specific study on solid nodules only is still missing.

For these reasons, the effectiveness of segmentectomy instead lobectomy for every kind of segment or tumor is still to be defined.

Aim of this study is to analyze survival outcome in patients underwent single or multiple segmentectomy compared to lobectomy in stage I non small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma or squamous cell carcinoma
* cStage cIA with or without nodal upstaging
* lymphoadenectomy
* age > 18 years old
* Radical resection
* anatomical resection (lobectomy or segmentectomy)
* PET CT done

Exclusion Criteria:

* Nodal or distant metastasis confirmed before surgery
* Pure solid GGO
* Follow up < 12 months
* Bilobectomy/pneumonectomy
* Trans fissure tumor
* Multiple lung tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected with NSCLC solid or part solid at the CT scan or PET CT study. These patients underwent anatomical resection with lymphoadenectomy and radical intent
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01-01; Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 1 YEAR
  Time between surgery and recurrence appearance

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Chiappetta, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Postmus PE, Kerr KM, Oudkerk M, Senan S, Waller DA, Vansteenkiste J, Escriu C, Peters S; ESMO Guidelines Committee. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv1-iv21. doi: 10.1093/annonc/mdx222. No abstract available. PMID 28881918
- [Background] Saji H, Okada M, Tsuboi M, Nakajima R, Suzuki K, Aokage K, Aoki T, Okami J, Yoshino I, Ito H, Okumura N, Yamaguchi M, Ikeda N, Wakabayashi M, Nakamura K, Fukuda H, Nakamura S, Mitsudomi T, Watanabe SI, Asamura H; West Japan Oncology Group and Japan Clinical Oncology Group. Segmentectomy versus lobectomy in small-sized peripheral non-small-cell lung cancer (JCOG0802/WJOG4607L): a multicentre, open-label, phase 3, randomised, controlled, non-inferiority trial. Lancet. 2022 Apr 23;399(10335):1607-1617. doi: 10.1016/S0140-6736(21)02333-3. PMID 35461558
- [Background] Okada M, Yoshikawa K, Hatta T, Tsubota N. Is segmentectomy with lymph node assessment an alternative to lobectomy for non-small cell lung cancer of 2 cm or smaller? Ann Thorac Surg. 2001 Mar;71(3):956-60; discussion 961. doi: 10.1016/s0003-4975(00)02223-2. PMID 11269480
- [Background] Schuchert MJ, Pettiford BL, Keeley S, D'Amato TA, Kilic A, Close J, Pennathur A, Santos R, Fernando HC, Landreneau JR, Luketich JD, Landreneau RJ. Anatomic segmentectomy in the treatment of stage I non-small cell lung cancer. Ann Thorac Surg. 2007 Sep;84(3):926-32; discussion 932-3. doi: 10.1016/j.athoracsur.2007.05.007. PMID 17720401
- [Background] Suzuki K, Saji H, Aokage K, Watanabe SI, Okada M, Mizusawa J, Nakajima R, Tsuboi M, Nakamura S, Nakamura K, Mitsudomi T, Asamura H; West Japan Oncology Group; Japan Clinical Oncology Group. Comparison of pulmonary segmentectomy and lobectomy: Safety results of a randomized trial. J Thorac Cardiovasc Surg. 2019 Sep;158(3):895-907. doi: 10.1016/j.jtcvs.2019.03.090. Epub 2019 Apr 9. PMID 31078312
- [Background] Wiley JL, Balster RL. Antipunishment activity of diazepam in rats trained to discriminate diazepam from vehicle. Exp Clin Psychopharmacol. 1999 Feb;7(1):13-9. PMID 10036605